CLINICAL TRIAL: NCT06213090
Title: Patterns of Disease, Outcomes and Treatment Response in Children With Neurodevelopmental Disorders
Brief Title: Patterns of Neurodevelopmental Disorders
Status: Recruiting | Type: Observational
Sponsor: Richard Frye (Other)
Collaborators: Autism Discovery and Treatment Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Richard Frye, Principal Investigator, Rossignol Medical Center
Organization: Rossignol Medical Center (Other)
Other Study IDs: NeuroClinical
Record Dates: First submitted 2024-01-04; First posted 2024-01-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Neurodevelopmental Disorders; Autism Spectrum Disorder; Pediatric Autoimmune Neuropsychiatric Disorder Associated With Streptococcal Infection; Pediatric Acute-Onset Neuropsychiatric Syndrome; Down Syndrome; Epilepsy; Mitochondrial Encephalomyopathies; Cerebral Folate Deficiency
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Pediatric acute-onset neuropsychiatric syndrome; Down Syndrome; Epilepsy; Mitochondrial Encephalomyopathies; Neurodegeneration Due To Cerebral Folate Transport Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, cerebrospinal fluid, muscle, and skin samples may be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Autism: Children with autism will be followed in regards to their clinical management.
- Mitochondrial Encephalopathy: Children with Mitochondrial Encephalopathy will be followed in regards to their clinical management.
- Down Syndrome: Children with Down Syndrome will be followed in regards to their clinical management.
- Cerebral Folate Deficiency: Children with Cerebral Folate Deficiency will be followed in regards to their clinical management.
- PANS: Children with PANS will be followed in regards to their clinical management.
- PANDAS: Children with PANDAS will be followed in regards to their clinical management.
- Epilepsy: Children with Epilepsy will be followed in regards to their clinical management.
- ADHD: Children with ADHD will be followed in regards to their clinical management.
- Dyslexia and other learning disabilities: Children with Dyslexia and other learning disabilities will be followed in regards to their clinical management.
- Other Neurodevelopmental Disorders: Children with Other Neurodevelopmental Disorders will be followed in regards to their clinical management.

SUMMARY:
The purpose of this study is to systematically evaluate the results of medical investigations to identify symptom and biological patterns and common etiologies of neurodevelopmental disorders.

DETAILED DESCRIPTION:
Although neurodevelopmental disorders are very prevalent (for example Autism affects 1 out of every 36 children and dyslexia affects up to 15% of the population), the etiology of such disorders is not known. The purpose of this investigation is to identify common etiologies of neurodevelopmental disorders (i.e., speech delay, global developmental delay, autism) and determine if it is possible to find early indicators of the diagnosis and foster the potential for a better prognosis of these disorders. At this time the investigators examine patients with neurodevelopment disorders with various medical investigations, but the results of these investigations are not systematically evaluated. One of the goals of this research is to systematically examine this information in order to identify patterns of test abnormalities that have not been previously described. Another goal of this research is to identify the common etiologies typically identified by the medical evaluation, so we can further refine our approach. In addition, the investigators now have the ability to evaluate biological samples for biomarkers that have potential to be diagnostically useful.

ELIGIBILITY:
Inclusion Criteria:

Neurodevelopmental delays Clinical visit at an Rossignol Medical Center

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who present to Rossignol Medical Center for standard care related to neurodevelopmental disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Specific Medical abnormalities | up to 7 years
  It is unknown if a specific set of biological abnormalities contribute to the formation of many types of neurodevelopmental disorders. The study is intended to identify the relationship between biological abnormalities and neurodevelopmental disorders. The chart will be reviewed for medical diagnoses other than the primary neurodevelopmental disorders.

SECONDARY OUTCOMES:
The number of children with abnormal clinical lab | up to 7 years
  It is unknown if a abnormalities in specific clinical laboratories are associated with specific neurodevelopmental disorders. The study is intended to identify the relationship between biological abnormalities and neurodevelopmental disorders. The medical chart will be reviewed to determine the number of children with a specific medical disorder who have abnormalities in specific clinical labs.
The number of children who respond to specific treatments | up to 7 years
  Various behavioral and medical treatments are used for many types of neurodevelopmental disorders but the effectiveness for many of these treatments is not known. The study is intended to identify the relationship between biological abnormalities (and their treatments) and neurodevelopmental disorders. The medical chart will be review to determine the treatments applied to each participant and the participants response.

CONTACTS AND LOCATIONS:
Locations (1):
- Rossignol Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified IPD may be shared on a case by case basis

REFERENCES:
- See also: Rossignol Medical Center — https://rossignolmedicalcenter.com/
- See also: Autism Discovery and Treatment Foundation — https://www.autismdiscovery.org/